CLINICAL TRIAL: NCT01285531
Title: Institutional Review Board Application #13373, Entitled "A Randomized Clinical Trial of Pediatric Lumbar Puncture Success Using The Compass, a Compact Quantitative Pressure Transducer
Brief Title: Pediatric Lumbar Puncture Success Using the COMPASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Life Sciences Development Fund (Unknown)
Responsible Party: Julie C. Brown, MD, MPH, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPASS13373
Record Dates: First submitted 2010-12-09; First posted 2011-01-28 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Lumbar Puncture
Keywords: lumbar puncture; Compass; pressure transducer; manometry; The focus of the study is to improve lumbar puncture(LP)success, reduce the number of LP attempts, reduce the number of traumatic attempts.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar puncture (No Intervention): The participants randomly assigned to this arm will receive a lumbar puncture using standard procedures and equipment
- Lumbar puncture with the Compass device (Experimental): The participants randomly assigned to this group will receive a lumbar puncture with the use of the Compass device.
  Interventions: Device: Compass Lumbar Puncture Enhanced

INTERVENTIONS:
Device: Compass Lumbar Puncture Enhanced — Participants randomly assigned to this group will receive a lumbar puncture using the Compass device.
  Other Names: compass
  Arms: Lumbar puncture with the Compass device

SUMMARY:
Objective: To evaluate pediatric emergency department provider lumbar puncture success with and without the Compass Lumbar Puncture Enhanced, a new pressure transducer, in order to determine: the proportion of lumbar punctures where a) any cerebrospinal fluid is obtained on the first attempt, b) any cerebrospinal fluid is obtained on any attempt, and c) sufficient cerebrospinal fluid is obtained for standard tests (culture, chemistries, cell count); the time to provider success in obtaining a) a drop of fluid from the needle, and b) opening pressure measurement; the proportion of successful lumbar punctures that contain blood; and provider satisfaction.

Background: Lumbar punctures are necessary to diagnose meningitis, neurological diseases and some cancers. They are common pediatric emergency department procedures that frequently require repeated attempts or are only partially successful, with sufficient blood to limit interpretation. Measuring cerebrospinal fluid pressure during lumbar punctures is recommended but rarely done, due to limitations of current technology. Liquid column manometry is cumbersome, time-consuming and frequently impractical. Existing pressure transduction probes that connect via tubing to external monitors are not designed or recommended for lumbar punctures. The pressure is displayed on a monitor that is difficult to view during the LP procedure and they equilibrate too slowly to keep pace of pressure changes during LPs. The Compass Lumbar Puncture Enhanced is a new, inexpensive, disposable, medical device, specifically designed for use during LPs, that has the potential to increase lumbar punctures success and decrease blood contamination. It attaches to the spinal needle and displays both a numeric pressure value and a pressure waveform, allowing physicians to more readily identify the cerebrospinal fluid space and measure cerebrospinal fluid pressure. The device is small, easy to use, and readily incorporated into standard practice.

The Compass Lumbar Puncture Enhanced uniquely provides immediate feedback about pressure that may allow physicians to more quickly and confidently identify the CSF space, and instantly determine cerebrospinal fluid pressure when the space is reached. The investigators believe the Compass Lumbar Puncture Enhanced will increase lumbar punctures success and decrease the proportion containing blood. It has the potential to become the standard of care and be used in every lumbar puncture procedure. This study is expected to demonstrate the clinical utility of the Compass Lumbar Puncture Enhanced to the medical community. Increased awareness of the Compass Lumbar Puncture Enhanced and a positive demonstration of the viability of the technology will help attract either the investment capital or the strategic partnership necessary to fully develop the market.

DETAILED DESCRIPTION:
Objective: To evaluate pediatric emergency department (ED) provider lumbar puncture success with and without the Compass Lumbar Puncture Enhanced, a new pressure transducer, in order to determine: the proportion of lumbar punctures (LPs) where a) any cerebrospinal fluid (CSF) is obtained on the first attempt, b) any CSF is obtained on any attempt, and c) sufficient CSF is obtained for standard tests (culture, chemistries, cell count); the time to provider success in obtaining a) a drop of fluid from the needle, and b) opening pressure measurement; the proportion of successful lumbar punctures that contain blood; and provider satisfaction.

Background: Lumbar punctures are necessary to diagnose meningitis, neurological diseases and some cancers. They are common pediatric emergency department procedures that frequently require repeated attempts or are only partially successful, with sufficient blood to limit interpretation. Measuring cerebrospinal fluid pressure during a lumbar puncture is recommended but rarely done, due to limitations of current technology. Liquid column manometry is cumbersome, time-consuming and frequently impractical. Existing pressure transduction probes that connect via tubing to external monitors are not designed or recommended for LPs. The pressure is displayed on a monitor that is difficult to view during the lumbar puncture procedure and they equilibrate too slowly to keep pace of pressure changes during lumbar puncture. The Compass Lumbar Puncture Enhanced is a new, inexpensive, disposable, medical device, specifically designed for use during lumbar punctures, that has the potential to increase lumbar puncture success and decrease blood contamination. It attaches to the spinal needle and displays both a numeric pressure value and a pressure waveform, allowing physicians to more readily identify the cerebrospinal fluid space and measure cerebrospinal fluid pressure. The device is small, easy to use, and readily incorporated into standard practice.

Methods: This randomized clinical trial will test adding the Compass Lumbar Puncture Enhanced vs. standard care in 60 children 0-16 years old who are receiving a lumbar puncture in the Seattle Children's Hospital Emergency Department. We will test the Compass Lumbar Puncture Enhanced against standard care in 60 children receiving lumbar puncture, comparing success, pressures obtaining, time to success, complications (e.g. >200 red blood cells/mm3) and provider satisfaction. Results will be compared with chi-squared tests, regressions, Kaplan-Meier and logrank tests. We expect improved success, decreased time to success and complications and high provider satisfaction.

Impact: Currently, one third of lumbar punctures require multiple attempts, 7-20% contain blood that limits interpretation, and 6% are unsuccessful. This results in unnecessary hospitalizations, increased hospital days, increased antibiotic use and increased numbers of repeat procedures. The Compass Lumbar Puncture Enhanced uniquely provides immediate feedback about pressure that will allow physicians to more quickly and confidently identify the cerebrospinal fluid space, and instantly determine cerebrospinal fluid pressure when the space is reached. We believe the Compass Lumbar Puncture Enhanced will increase lumbar puncture success and decrease the proportion containing blood. It has the potential to become the standard of care and be used in every lumbar puncture procedure. This study is expected to demonstrate the clinical utility of the Compass Lumbar Puncture Enhanced to the medical community.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 - 18 years old
* Patient was in the Seattle Children's Hospital (SCH) Emergency Department (ED)within 24 hours
* Patient requires lumbar puncture (can be performed in the ED or inpatient, within 24 hours of arrival to the ED)
* Parent is able to read English or Spanish
* A provider who is trained in the use of the Compass device is willing and able to use it during the LP

Exclusion Criteria:

* Child is a foster child or ward of the state or is unaccompanied by their legal guardian
* Child has a lower spine deformity, such as spina bifida, that would impact lP success
* The child is pregnant, by verbal report or clinically available test results

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Lumbar puncture success | 1 minute to 2 hours
  Time to lumbar puncture success. In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine the proportion of LPs where any CSF is obtained on any attempt

SECONDARY OUTCOMES:
Obtaining CSF fluid | 1 minute to 2 hours
  In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine the proportion of LPs where any CSF is obtained on any attempt
Obtain sufficient CSF fluid | 1 minute to 2 hours
  In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine the proportion of LPs where sufficient CSF is obtained for standard tests (culture, chemistries and cell count) on any attempt
Successful traumatic LPs (contaminated with blood) | 1 minute to 2 hours
  In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine the proportion of successful LPs that are traumatic (contaminated with blood)
Time to fluid | 1 minute to 2 hours
  In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine the time to provider success in obtaining a drop of fluid from the needle
Time to LP opening pressure | 1 minute to 2 hours
  In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine the time to provider success in obtaining opening pressure measurement
Provider satisfaction | 1 minute to 2 hours
  In pediatric patients receiving emergency department care, we aim to evaluate pediatric ED provider LP success with and without the Compass, in order to determine provider satisfaction with the procedure +/- device.

CONTACTS AND LOCATIONS:
Overall Officials: JUlie C. Brown, MD, MPH, Principal Investigator — Seattle Children's Hospital, Pediatric Emergency Department
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States